CLINICAL TRIAL: NCT03634748
Title: Thrombolysis in stRoke With Unknown onSet Based on Non-contrasT CT (TRUST CT). An International, Multicenter, Registry-based Study
Brief Title: Thrombolysis in stRoke With Unknown onSet Based on noncontrasT CT
Acronym: TRUST CT
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: St John of God Hospital, Vienna (Other)
Responsible Party: Principal Investigator, Dr. Sven Poli, Deputy Director, University Hospital Tuebingen
Other Study IDs: TRUST CT
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicentric, observational, registry-based study of 0.9 mg/kg i.v. thrombolysis in wake-up stroke or stroke with unknown onset based on non-contrast CT appearance only

DETAILED DESCRIPTION:
Thrombolysis in wake-up stroke (WUS) or stroke with unknown onset (SUO) has been recently proven to be safe and effective using magnetic resonance imaging (MRI). However, in most of the thrombolyzing hospitals worldwide MR imaging is not available. We hypothesize that pragmatic non-contrast CT (NCCT)-based WUS/SUO thrombolysis may be feasible and safe.

Methods: TRUST-CT is an international multicenter registry-based study. WUS/SUO patients undergoing NCCT-based thrombolysis with NIHSS ≥ 4 and initial ASPECTS ≥ 7 are included and compared to propensity score matched non-thrombolyzed WUS/SUO controls. Primary endpoint is symptomatic intracranial hemorrhage (ICH); secondary endpoints include 24-hour NIHSS change of ≥ 4 and modified Rankin Score (mRS) at 90 days.

ELIGIBILITY:
Inclusion:

1. Ischemic stroke with NIHSS ≥ 4
2. Wake-up stroke or unknown onset stroke
3. Age ≥ 18 years
4. rtPA Bolus within 4.5h of awakening and/or within 4.5 of discovering symptoms
5. rtPA Bolus within 30 min. of admission CT

Exclusion:

1. Noncontrast cranial CT scan with ASPECTS < 7
2. Evidence of intracranial or subarachnoid hemorrhage
3. Inability to control systolic BP >185mm Hg, or diastolic BP >110mm Hg with IV antihypertensive medication
4. Known coagulopathy or evidence of active bleeding
5. Surgical procedures, subclavian arterial puncture, trauma, and gastrointestinal or genitourinary bleeding within 14 days of the event
6. Patients taking oral anticoagulants and having an INR >1.7
7. A platelet count <100 000, venous glucose either <50 or >450
8. Premorbid mRS > 3

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: wake-up stroke, unknown onset stroke
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
sICH | 72hours
  symptomatic ICH according to ECASS3

SECONDARY OUTCOMES:
mRS 90 days | 90 days
  mRS 90 days

CONTACTS AND LOCATIONS:
Locations (5):
- St. Johns Hospital Vienna, Vienna, Austria
- University Hospital Tuebingen, Tübingen, Germany
- Slovakia (2):
  - University Hospital Bratislava, Bratislava
  - General Hospital Liptovsky Mikulas, Liptovský Mikuláš
- Lausanne University Hospital, Lausanne, Switzerland

REFERENCES:
- [Derived] Sykora M, Kellert L, Michel P, Eskandari A, Feil K, Remi J, Ferrari J, Krebs S, Lang W, Serles W, Siarnik P, Turcani P, Kovacik M, Bender B, Mengel A, Poli K, Poli S. Thrombolysis in Stroke With Unknown Onset Based on Non-Contrast Computerized Tomography (TRUST CT). J Am Heart Assoc. 2020 Feb 18;9(4):e014265. doi: 10.1161/JAHA.119.014265. Epub 2020 Feb 12. PMID 32067594